CLINICAL TRIAL: NCT05272943
Title: Oxygen Saturation Measurement With Pulse Oximetry and Smart Phones and Smart Wearable: Prospective Observational Trial
Brief Title: Oxygen Saturation Measurement With Pulse Oximetry and With Smart Phones and Smart Wearable
Acronym: SATURATE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Other Study IDs: KDAR SATURATE 2022
Record Dates: First submitted 2022-02-17; First posted 2022-03-10 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Oxygen Saturation Measurement
Keywords: pulse oximetry; pediatric patient; smart phone; smart wearable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Preanesthesia visit measurement: Oxygen saturation will be measured by validated pulse oxymetry and smart electronics in pediatric patients during preanesthesia visit
  Interventions: Other: Oxgen saturation measurement with validated pulse oximetry; Other: Oxgen saturation measurement with smart electronics
- General anesthesia measurement: Oxygen saturation will be measured by validated pulse oxymetry and smart electronics in pediatric patients during general anesthesia
  Interventions: Other: Oxgen saturation measurement with validated pulse oximetry; Other: Oxgen saturation measurement with smart electronics
- PACU measurement: Oxygen saturation will be measured by validated pulse oxymetry and smart electronics in pediatric patients during PACU stay
  Interventions: Other: Oxgen saturation measurement with validated pulse oximetry; Other: Oxgen saturation measurement with smart electronics
- PICU measurement: Oxygen saturation will be measured by validated pulse oxymetry and smart electronics in pediatric patients during PICU stay
  Interventions: Other: Oxgen saturation measurement with validated pulse oximetry; Other: Oxgen saturation measurement with smart electronics

INTERVENTIONS:
Other: Oxgen saturation measurement with validated pulse oximetry — Oxgen saturation will be measured with validated pulse oximetry
Other: Oxgen saturation measurement with smart electronics — Oxgen saturation will be measured with smart electronics

SUMMARY:
Oxgen saturation measurement with the pulse oximetry is considered as a standard of care for respiratory system monitoring. The evaluation of measured oxygen saturation could lead to the clinical decision making in taking care of patient with respiratory failure. Smart electronics (such smart phones, smart watch, and others) are currently equipped with the sensors and applications that allows the peripheral oxygen saturation, however the corelation between the validated measurement (pulse oximetry) and smart electronics measurement is not known at the moment. In case of close correlation and high sensitivity, could be the smart electronics used for oxygenation evaluation of outpatients together with possible early deterioration detection.

DETAILED DESCRIPTION:
After informed consent from patients and/or legal guardian the oxygen saturation will be measured by calibrated pulse oxymetry (validated for medical use only) and by smart electronics (smart phones and smart wearable) in pediatric patients during the preanesthesia evaluation, under general anesthesia, during the postanesthesia care unit (PACU) stay, and at pediatric intensive care unit (PICU) stay. In one patient, overall 6 measurements in will be performed (3 on right and 3 on left hand).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* pediatric patients during preanesthesia visit
* pediatric patients during general anesthesia
* pediatric patients during PACU stay
* pediatric patients during PICU stay

Exclusion Criteria:

* outside age limits
* refused to participate

Ages: 1 Year to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric patients during during preanesthesia visit, general anesthesia, PACU and PICU stay will be eligible for inclusion
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Pulse oximetry correlation | Perioperatively
  Pulse oximetry correlation between the validated pulse oximetry and smart electronics

SECONDARY OUTCOMES:
Measurement tolerance | Perioperatively
  The tolerance of measurement will be evaluated by number of valid measurement attempts

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, prof. MD., Ph.D., MBA, Study Chair — Department of paediatric anaesthesia and intensive care medicine
Locations (1):
- Brno University Hospital, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided